CLINICAL TRIAL: NCT03328481
Title: Quadratus Lumborum Block Using Loss-of-resistance Versus Ultrasound-guided Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N-88-2017
Record Dates: First submitted 2017-10-29; First posted 2017-11-01 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Lower Abdominal Surgery; Quadratus Lumborum Block
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Loss-of-resistance (Experimental): Patients in this group will receive Loss-of-resistance Quadratus lumborum block with 30 ml bupivacaine 0.25% in addition to general anesthesia.
  Interventions: Procedure: Loss-of-resistance Quadratus lumborum block; Procedure: General anesthesia
- Ultrasound-guided (Active Comparator): Patients in this group will receive Ultrasound-guided Quadratus lumborum block type-II with 30 ml bupivacaine 0.25% in addition to general anesthesia.
  Interventions: Procedure: Ultrasound-guided Quadratus lumborum block; Procedure: General anesthesia

INTERVENTIONS:
Procedure: Loss-of-resistance Quadratus lumborum block — ِA blunted 22-G, 11 mm, short-bevel facet needle will be introduced in the paravertebral line at the level of L3 or L4, in 30-45 degree to the skin directing it laterally. Once the skin barrier is breached, the needle will be withdrawn back so that the tip lies just under the skin. The needle will be advanced through the posterior thoracolumbar fascia and a first fast "pop" sensation will be felt when the needle pierced it. With further advancement of the needle, a second deep pop will be felt after it pierces the middle thoracolumbar fascia. At this point, the needle will be in the plane of the quadratus lumborum block type II. After careful aspiration, the 30 mLs of local anaesthetic will be injected. The needle will be visualized by the ultrasound by another physician to ensure safety.
  Arms: Loss-of-resistance
Procedure: Ultrasound-guided Quadratus lumborum block — A broadband (5-8 MHz) convex transducer will be placed transversely in the abdominal flank above the iliac crest to identify the external oblique, internal oblique, transversus abdominis muscles and aponeurosis. Then the external oblique muscle will be followed posteriorly until its posterior border is visualized (hook sign), and the posterior aspect of the Quadratus lumborum muscle is confirmed. A 22-G, 11-mm, short-bevel facet needle will be advanced under direct ultrasound visualization in-plane from anterolateral to postero-medial. Then the 30 ml of local anesthetic (bupivacaine 0.25 %) will be injected into the lumbar inter-facial triangle (LIFT) behind the quadratus lumborum muscle using hydro-dissection.
  Arms: Ultrasound-guided
Procedure: General anesthesia — Patients will receive 2 mg of midazolam and 8 mg of dexamethasone IV; then, they will be transferred to the operating room to receive a standard general anesthetic. Perioperative monitoring will include ECG, non-invasive arterial blood pressure, and pulse oximetry (SpO2) and end-tidal carbon dioxide. Anesthesia will be induced by propofol 1.5-2.5 mg/kg, atracurium 0.5 mg/kg, and fentanyl 2 mcg/kg to facilitate the insertion of an endotracheal tube. Anesthesia will be maintained by isoflurane 1-2% end-tidal concentration to maintain systolic arterial blood pressure and heart rate within + 20% of the baseline values. Ventilation will be adjusted to maintain normocapnia.

SUMMARY:
This study aims to explore the feasibility of using loss-of-resistance technique for Quadratus Lumborum block (QLB). And to compare between the Ultrasound guided QLB type II and the loss-of-resistance technique for QLB as regards the degree and duration of analgesia and side effects.

DETAILED DESCRIPTION:
Quadratus lumborum block (QLB) is an abdominal plane block with increasing popularity. QLB is achieved by local anesthetic infiltration at the anterolateral aspect of quadratus lumborum muscle (QLB-I), or at the posterior aspect of the muscle (QLB-II), or transmuscular (QL-TM block). Ultrasound-guided technique is the usual route used for QLB performance. QLB had been considered a modification of transversus abdominis plane (TAP) block[4]. A cadaveric study had showed similar local anesthetic spread in both QL and TAP blocks.

TAP block could be performed by using either the ultrasound or loss-of-resistance technique; whilst, QLB is only performed using the ultrasound and the feasibility of loss-of-resistance technique had not been investigated for this block.

This study aims to explore the feasibility of using loss-of-resistance technique for QLB. And to compare between the Ultrasound guided QLB type II and the loss-of-resistance technique for QLB as regards the degree and duration of analgesia and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for lower abdominal surgery under general anesthesia

Exclusion Criteria:

* Patient refusal to regional block,
* Pregnancy
* Coagulopathy
* Cognitive impairment
* Inflammation or infection at the puncture site
* History of allergic reaction to study medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2018-05-28 (Actual); Primary Completion 2018-09-15 (Estimated); Study Completion 2018-09-20 (Estimated)

PRIMARY OUTCOMES:
Duration of analgesia | 24 hours
  The time between the end of the surgery and the first analgesia request

SECONDARY OUTCOMES:
Postoperative morphine consumption | 24 hours
  The total amount of morphine needed during the first 24 hours
Intraoperative extra-analgesia requirements | 3 hours
  The total amount of analgesic drug boluses
visual analogue pain score at rest to assess the pain severity | 24 hours
  the grade of pain experienced by the patient at rest graded from 0 to 10. The lower the value, the better the score
Visual analogue pain score at movement to assess the pain severity | 24 hours
  the grade of pain experienced by the patient at movement graded from 0 to 10. The lower the value, the better the score
Systolic blood pressure | 24 hours
  the systolic blood pressure measured in mmHg
Heart rate | 24 hours
  The number of heart beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Mukhtar, Study Director — Head of research committee section in anesthesia department
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No